CLINICAL TRIAL: NCT00737763
Title: Beta Cell Rescue in New Onset Type 1 Diabetes Mellitus With the LFA-1 Antibody Efalizumab
Brief Title: Beta Cell Rescue in New Onset Type 1 Diabetes With Efalizumab
Acronym: BRiTE
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: drug withdrawn from market
Sponsor: Emory University (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other); Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Mark Rigby, Principal Investigator, Emory University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB0007365; BRiTE Trial for T1DM (Other: Other)
Record Dates: First submitted 2008-08-19; First posted 2008-08-20 (Estimated); Last update posted 2014-05-12 (Estimated); Status verified 2014-05

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: efalizumab; Raptiva; Diabetes; Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus | interventions — efalizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): This group will receive weekly efalizumab injections for 6 months
  Interventions: Drug: efalizumab
- B (Placebo Comparator): This group will receive placebo injections for 6 months
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: efalizumab — Enrollees randomized to efalizumab will receive the first dose of 0.7mg/kg subcutaneously given at enrollment, and 1.0 mg/kg subcutaneously weekly for 26 weeks self or family-administered after injection training. This is the FDA-approved initial and subsequent doses of efalizumab used for psoriasis treatment
  Other Names: Raptiva
  Arms: A
Drug: placebo — Enrollees receiving placebo will be given a subcutaneous injection of equal volume and appearance to treatment on the same schedule.
  Other Names: none applicable
  Arms: B

SUMMARY:
In this single-center therapeutic study, we will study the ability of efalizumab to protect remaining beta cells in teenagers and young adults who have been newly diagnosed with type 1 diabetes mellitus. Efalizumab is a monoclonal antibody which prevents the activation of antigen specific T lymphocytes to sites of inflammation. Efalizumab was approved by the FDA in 2003 for the treatment of psoriasis. It has been proven to be safe, well tolerated and effective in targeting T cell mediated disorders like those seen in autoimmunity.

DETAILED DESCRIPTION:
Since there is data that shows that early intervention can prevent further destruction of insulin producing beta cells, the patients who will be enrolled in this study will have been diagnosed with Type 1 diabetes within 6 weeks of enrolling and starting therapy. Patients who meet the screening criteria will be randomized at a 2 to 1 ratio to either get weekly subcutaneous injections of efalizumab for 26 weeks versus a placebo injection. The researchers and patients will be blinded to the treatment group assignment. All patients will be followed for two years.

The primary endpoint for this study will be the difference from baseline in the body's ability to respond to a Mixed Meal Tolerance Test at 12 months after enrollment. The Mixed Meal Tolerance test will help test the production of insulin by the pancreas. By comparing the results of these tests between the treated group and the placebo group, we hope to be able to show preservation of beta cell function in the group treated with efalizumab.

ELIGIBILITY:
Inclusion Criteria:

* Males or females 12-35 years old, no preference nor discrimination will be made based on ethnicity.
* Recent diagnosis of Type 1Diabetes Mellitus, participant can be enrolled in the trial within 6 weeks of diagnosis.
* Positive for at least one diabetes autoantibody. Insulin autoantibody positivity will only be used as a selection criterion if insulin has not been used in at least the preceding 10 days.
* Willingness to provide written informed consent (either the subject or the subject's legally authorized representative)
* Have routine diabetic care under an endocrinologist and ability to follow study protocol for the duration of the 2-year study.
* Although no preference or discrimination will be made based on ethnicity or gender, participants (and family and/or guardians when applicable) must demonstrate comprehension of the trial, including its obligations and potential risks.
* If a female of childbearing potential, a negative pregnancy test and commitment to the use of two forms of effective contraception or abstinence for the duration of the study are necessary.
* If a non-sterile male, commitment to the use of two forms of effective contraception (birth control) for the duration of the study is necessary.

Exclusion Criteria:

* Severe allergic allergy or anaphylaxis to human monoclonal antibodies
* Hospital admission for cardiac disease, stroke, or pulmonary disease within the past year
* History of substance abuse within last 5 years
* History of ongoing uncontrolled bacterial, viral, or fungal or atypical mycobacterium infections
* History of opportunistic infections
* Diagnosis with hepatic cirrhosis regardless of cause or severity
* Diagnosis, history, or laboratory evidence of Hepatitis B or C infection
* Hepatic enzymes 2 > times the upper limit of normal
* History of active or treatment for tuberculosis or skin test positive
* History of malignancy over the past 5 years
* Recent initiation or change in treatment regimen of beta-blockers, angiotensin-converting enzyme inhibitors, interferons, quinidine anti-malarial drugs, or lithium in the past month
* Seropositivity for human immunodeficiency virus (HIV)
* Serologic or clinical evidence of recent or acute infection with Epstein-Barr Virus or Cytomegalovirus
* Females who are pregnant, lactating, or planning on pregnancy during the 2 year study period
* Progressive hearing loss
* History of organ or bone marrow transplantation, sickle cell disease, cystic fibrosis, autoimmune anemia, seizures, autoimmune thrombocytopenia, leuko/lymphopenia, vasculitis, other autoimmune disease.
* Current use of immunosuppressive medications
* Plan or requirement of receiving new immunization of any type within the first 12 months of the study, or booster or completion vaccines with live or live-attenuated vaccines
* Any condition that, in judgment of the investigator, could jeopardize the subject-safety following exposure to the drug.
* Participation in another simultaneous medical investigation or trial

Ages: 12 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2008-10; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
The primary endpoint for this study will be the difference from baseline in the body's ability to respond to a Mixed Meal Tolerance Test at 12 months after enrollment. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Mark R Rigby, MD, PhD, Principal Investigator — Emory University, Children's Healthcare of Atlanta; Eric Felner, MD, Principal Investigator — Children's Healthcare of Atlanta, Emory University; Sol Jacobs, MD, Principal Investigator — Emory University; Christian Larsen, MD, DPhil, Principal Investigator — Emory University